CLINICAL TRIAL: NCT02027844
Title: Cartoon Distraction and Parental Presence During Induction of Anesthesia on Preoperative Anxiety and Postoperative Behavior Change in Children Undergoing General Anesthesia
Brief Title: Cartoon Distraction and Parental Presence on Anxiety in Pediatric Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sung Mee Jung, Associate professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JUNG999ANXIETY
Record Dates: First submitted 2013-12-30; First posted 2014-01-06 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Anxiety, Separation; Psychomotor Agitation
MeSH Terms: conditions — Anxiety, Separation; Psychomotor Agitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cartoon (Experimental): cartoon watching by children during inhalational induction of anesthesia in the operating room
  Interventions: Behavioral: Cartoon
- Paretnal presence (Active Comparator): parental presence with their children during inhalational induction of anesthesia in the operating room
  Interventions: Behavioral: parental presence
- Combined (Experimental): parental presence and cartoon watching by children during inhalational induction of anesthesia in the operating room
  Interventions: Behavioral: Cartoon; Behavioral: parental presence

INTERVENTIONS:
Behavioral: Cartoon — Cartoon watching by children during inhalational induction of sevoflurane
  Other Names: Cartoon watching by children
  Arms: Cartoon; Combined
Behavioral: parental presence — parental presence during inhalational induction of sevoflurane
  Arms: Combined; Paretnal presence

SUMMARY:
Nearly 50% of young children undergoing surgery exhibit high level of anxiety during induction of anesthesia because of exposure to unfamiliar environment and people and separation from parents. Increased preoperative anxiety may impact postoperative behavior changes such as emergence agitation, separation anxiety and sleep disturbance. Although some pediatric anesthesiologists routinely permit parental presence to reduce the anxiety during induction of anesthesia, previous studies have reported conflicting results. Recently the distraction using video game or animated cartoon has been reported to reduce anxiety of young children during induction of anesthesia. However, it was still undetermined whether distraction has its own ability to reduce children's anxiety separated from parental presence because they evaluated the effect of video method in the parental presence. The investigators design to investigated the efficacy of distraction with watching cartoon, parental presence and combined with watching cartoon and parental presence on reduction of anxiety during inhalational induction of anesthesia using sevoflurane. In addition this study includes long-term effect of each intervention such as postoperative emergence agitation and postoperative behavior change in children.

DETAILED DESCRIPTION:
This study is different from previous reports as follow. First, investigators separate the effect of cartoon distraction and parental presence on minimizing preoperative anxiety and determine whether an interaction between two different interventions is existent. Second, investigators evaluate the effect of preoperative anxiety on the long-term behavioral change of children. It was not clarified yet in clinical practice. Third, investigators evaluate the effect of each intervention on parental anxiety before and after induction of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status 1 and 2
2. 1-7 years old.
3. elective, single minor surgery under general anesthesia

Exclusion Criteria:

1.Chronic illness, psychological or emotional disorder, abnormal cognitive development 2.Previous anesthetic experience 3.Closure both eyes after surgery 4.Sedative medication or psychoactive drugs medication, 5.History of allergy to the drugs used in our study 6.Expected difficult intubation or respiration such as abnormal airway, reactive airway disease, upper respiratory infection in recent 3 weeks

-

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Mee Jung, MD, Principal Investigator — Yeungnam University College of Medicine
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

REFERENCES:
- See also: Streamed video clips to reduce anxiety in children during inhaled induction of anesthesia — http://www.ncbi.nlm.nih.gov/pubmed/23051880
- See also: Cartoon distraction alleviates anxiety in children during induction of anesthesia — http://www.ncbi.nlm.nih.gov/pubmed/23011563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted Yeungnam University Hospital in South korea from Dec. 30. 2013 to October. 31. 2014. One hundred and seventeen children aged between 2 and 7 years, ASA physical status I or II scheduled for elective minor surgery under general anesthesia were enrolled. .
Pre-assignment Details: Children with a chronic illness, developmental delay, a neuropsychiatric disease, cancer, experience of a recent stressful life event, previous anesthetic experience, sedative medication, or emergency surgery were excluded.
Period: Overall Study
Arm/Group | Cartoon | Paretnal Presence | Combined
Started | 39 | 39 | 39
Completed | 34 | 33 | 37
Not Completed | 5 | 6 | 2
Not completed — Withdrawal by Subject | 3 | 2 | 1
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — Incomlete data | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cartoon | Paretnal Presence | Combined | Total
Number analyzed (Participants) | 34 | 33 | 37 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 33 | 37 | 104
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.5 (1.0) | 5.3 (1.4) | 5.0 (1.3) | 5.2 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 19 | 59
  Male | 15 | 12 | 18 | 45

OUTCOME MEASURES:

1. Primary Outcome: Modified Yale Preoperative Anxiety Scale Scores at Baseline, Arrival in Operating Room, and Inhalation Induction
Description: The investigators measure change in anxiety of children using Modified Yale Preoperative Anxiety scale (m-YPAS): Scale changes from Activities, Vocalization, Expressing emotions, State of arousal, Interaction with family members.
  Each domain received a partial score based on the punctuation observed divided by the number of categories of that domain. The score of each domain is added to the others
  Total scores ranged from 23.4 to 100 The scores considered "cut points" to determine whether a patient had/had not anxiety were 23
  * Without anxiety: 23.4 e 30
  * With anxiety: greater than 30.
Time Frame: 1. baseline (10 minute after arrival in the preoperative holding area) 2. on arrival in the operating room, 3. during inhalational induction with sevoflurane
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Cartoon | Paretnal Presence | Combined
Number analyzed (Participants) | 34 | 33 | 37
units on a scale
  Preoperative holding area | 28.4 [23.4 to 36.6] | 28.4 [23.4 to 46.6] | 23.4 [23.4 to 65.3]
  Entrance to the operating room | 23.4 [23.4 to 31.6] | 33.4 [23.4 to 50.0] | 28.4 [23.4 to 46.6]
  Induction | 28.4 [23.4 to 46.6] | 43.4 [23.4 to 65.0] | 43.4 [23.4 to 70.0]

2. Secondary Outcome: Change From Baseline Parental Anxiety at Postinduction of Anesthesia
Description: The investigators measure change of parental anxiety using State-Trait Anxiety Inventory (STAI)
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory and consists of 40 questions on a self-report basis.
  The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic.
  Higher scores are positively correlated with higher levels of anxiety.
  Each type of anxiety has its own scale of 20 different questions that are scored.
  Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Time Frame: 1. baseline: 15 minute after arrival at preoperative holding area before induction of anesthesia 2. postinduction : after induction of anesthesia
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Cartoon | Paretnal Presence | Combined
Number analyzed (Participants) | 34 | 33 | 37
units on a scale | 0.0 [-6.0 to 3.0] | 0.0 [-3.0 to 3.0] | 0.0 [0.0 to 3.0]

3. Other Pre Specified Outcome: Postoperative Emergence Delirium
Description: The investigators measure postoperative emergence delirium of children after recovery of anesthesia using Children's Hospital of Eastern Ontario Pain(CHEOP) Scale at 20 minute in postanesthetic care unit
  The CHEOPS (Children's Hospital of Eastern Ontario Pain Scale) is a behavioral scale for evaluating postoperative pain in young children. It can be used to monitor the effectiveness of interventions for reducing the pain and discomfort.
  CHEOPS pain score = SUM(points for all 6 parameters) : Cry, facila, Child verbal, Torso, Touch, legs
  Interpretation:
  * minimum score: 4 = no pain
  * maximum score: 13 = the worst pain
  When the highest CHEOPS score recorded at any time exceeded 10, emergence delirium was deemed to be present.
Time Frame: at 20 minute in postanesthetic care unit
Population: When the highest CHEOPS score recorded at any time exceeded 10, emergence delirium was deemed to be present.
Measure: Number; unit: participants
Arm/Group | Cartoon | Paretnal Presence | Combined
Number analyzed (Participants) | 34 | 33 | 37
participants | 13 | 13 | 20

4. Other Pre Specified Outcome: Postoperative Behavioral Changes
Description: The investigators measure negative postoperative behavioral change of children after discharge of postanesthetic care unit using posthospital behavioral questionnaires( PHBQ ) at postoperative day (POD) 1 by visiting and followed at POD 14 by phone interview.
  The PHBQ consists of 27 items concerning sleep, eating, anxiety, aggressive behaviour, etc.
  The subscales were: general anxiety and regression, separation anxiety, anxiety about sleep, eating disturbance, aggression towards authority, and withdrawal.
  Negative behavior change was evaluated in 6 subscales categories. If more than one negative behavior change developed, the investigators calculated number of children who developed new-onset negative behavior change.
Time Frame: 1. postoperative 2 days, 2 postoperative 14 days
Population: If more than one negative behavior change in children developed, the investigators calculated number of the children who developed new-onset negative behavior change.
Measure: Number; unit: participants
Arm/Group | Cartoon | Paretnal Presence | Combined
Number analyzed (Participants) | 34 | 33 | 37
participants
  postoperative 2 days | 17 | 19 | 15
  postoperative 14 days | 7 | 5 | 3

ADVERSE EVENTS:
Arm/Group | Cartoon | Paretnal Presence | Combined
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/37
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/37

LIMITATIONS AND CAVEATS:
Parental anxiety was assessed using a self-reporting rating scale. we did't measure the baseline temperament of children using a validated behavioral assessment tool and were unable to calculate the 'use of parents' item of the mYPAS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No